CLINICAL TRIAL: NCT00164749
Title: A Pilot Study of Curcumin and Ginkgo for Treating Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: BUPA Foundation (Other); Kwong Wah Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE-2003.090-T
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Alzheimer's Disease
Keywords: dementia; cognition; memory; neurodegenerative disease; brain
MeSH Terms: conditions — Alzheimer Disease; Dementia; Neurodegenerative Diseases | interventions — Ginkgo Extract; Curcumin

ARMS (3):
- Placebo (Placebo Comparator): Color-matched placebo
  Interventions: Drug: Placebo and ginkgo extract
- 1 gram (Experimental): 1 g/day curcumin
  Interventions: Drug: Curcumin and ginkgo extract
- 4 gram (Experimental): 4 g/day curcumin
  Interventions: Drug: Curcumin and ginkgo extract

INTERVENTIONS:
Drug: Placebo and ginkgo extract — Placebo once daily, either as capsules or as powder to be mixed with food. All patients also received 120 mg/day standardized ginkgo leaf extract.
  Arms: Placebo
Drug: Curcumin and ginkgo extract — 1 g curcumin once daily, either as capsules or as powder to be mixed with food. All patients also received 120 mg/day standardized ginkgo leaf extract.
  Arms: 1 gram
Drug: Curcumin and ginkgo extract — 4 g curcumin once daily, either as capsules or as powder to be mixed with food. All patients also received 120 mg/day standardized ginkgo leaf extract.
  Arms: 4 gram

SUMMARY:
The purpose of this study is to develop procedures for testing the effectiveness of curcumin on slowing Alzheimer's disease (AD) progression.

DETAILED DESCRIPTION:
A double-blind, randomized, clinical trial of 30 subjects will be carried out to develop procedures for testing the effectiveness of curcumin on slowing Alzheimer's disease (AD) progression. Curcumin is a polyphenolic molecule extracted from turmeric and is widely and safely used as a yellow food coloring. Because of its strong anti-inflammatory activity, curcumin was tested in animal models of AD, where it significantly reduced levels of brain amyloid, oxidized proteins, and isoprostanes, and prevented cognitive deficits. AD patients will receive placebo, 1 g, or 4 g of curcumin daily for six months. All patients will also receive 120 mg ginkgo leaf extract daily. At 0, 1, 3, and 6 months of the study, a cognitive test will be performed, and blood samples will be analyzed for levels of isoprostane, amyloid beta protein, metals, and cholesterol. Curcumin and its metabolites will be measured in blood at 1 month. The primary objective for this first human study of curcumin in AD is to examine safety and procedures for a possible larger trial testing curcumin against AD. The secondary objective is to determine whether curcumin affects biochemical measures, and, if so, which dose is most effective. The tertiary objective is to determine whether curcumin slows cognitive decline in AD. This study may lead to inexpensive treatment that delays progression of AD.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic Chinese living in Hong Kong
* Progressive decline in memory and cognitive function for at least 6 months
* NINCDS-ADRDA diagnosis of possible or probable AD
* Mild to severe dementia with Cantonese version of MMSE scores between 0 and 28
* Informed consent from patient and/or caregiver
* Both elderly home residents and outpatients are eligible
* Patients may take any medication

Exclusion Criteria:

* Anticoagulant or antiplatelet treatment or bleeding risk factors
* Currently smoking
* Other severe, end-stage illness

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Change in isoprostane level in plasma | 1 and 6 months
Change in A-beta level in serum | 1 and 6 months

SECONDARY OUTCOMES:
Change in cognitive function (MMSE score) | 6 months
Change in cholesterol and triglycerides in serum | 1 and 6 months
Change in metals in serum | 1 month
Level of curcumin in plasma vs. dose | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Larry Baum, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

REFERENCES:
- [Result] Baum L, Lam CW, Cheung SK, Kwok T, Lui V, Tsoh J, Lam L, Leung V, Hui E, Ng C, Woo J, Chiu HF, Goggins WB, Zee BC, Cheng KF, Fong CY, Wong A, Mok H, Chow MS, Ho PC, Ip SP, Ho CS, Yu XW, Lai CY, Chan MH, Szeto S, Chan IH, Mok V. Six-month randomized, placebo-controlled, double-blind, pilot clinical trial of curcumin in patients with Alzheimer disease. J Clin Psychopharmacol. 2008 Feb;28(1):110-3. doi: 10.1097/jcp.0b013e318160862c. No abstract available. PMID 18204357
- [Result] Baum L, Cheung SK, Mok VC, Lam LC, Leung VP, Hui E, Ng CC, Chow M, Ho PC, Lam S, Woo J, Chiu HF, Goggins W, Zee B, Wong A, Mok H, Cheng WK, Fong C, Lee JS, Chan MH, Szeto SS, Lui VW, Tsoh J, Kwok TC, Chan IH, Lam CW. Curcumin effects on blood lipid profile in a 6-month human study. Pharmacol Res. 2007 Dec;56(6):509-14. doi: 10.1016/j.phrs.2007.09.013. Epub 2007 Sep 18. PMID 17951067